CLINICAL TRIAL: NCT03190174
Title: A Phase 1/2 Study Using Nivolumab and ABI-009 for Advanced Sarcoma, Advanced Carcinoma Treated With PD1 Inhibitors, and Tumors With Genetic Mutations Sensitive to mTOR Inhibitors
Brief Title: Nivolumab (Opdivo®) Plus ABI-009 (Nab-rapamycin) for Advanced Sarcoma and Certain Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-1701
Record Dates: First submitted 2017-02-02; First posted 2017-06-16 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Ewing Sarcoma; PEComa; Epithelioid Sarcoma; Desmoid Tumor; Chordoma; Non Small Cell Lung Cancer; Urothelial Carcinoma; Melanoma; Renal Cell Carcinoma; Squamous Cell Carcinoma; Hepatocellular Carcinoma; Classical Hodgkin Lymphoma; Colorectal Cancer; MTOR Activating Mutation
MeSH Terms: conditions — Sarcoma, Ewing; Perivascular Epithelioid Cell Neoplasms; Sarcoma; Desmoid Tumors; Chordoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Melanoma; Carcinoma, Renal Cell; Carcinoma, Squamous Cell; Carcinoma, Hepatocellular; Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): This is an open label, dose-seeking phase 1b study using a defined dose of nivolumab and escalating doses of Nab-Rapamycin (ABI-009) given intravenously.
  I. Dose Escalation Phase 1 Part of Study: The study will employ the standard "cohort of three" design. No intra-patient dose escalation will take place.
  II. Expansion Phase 1b Part of Study: Following dose escalation, an additional 22-28 patients will receive ABI-009 at the MTD and defined doses of nivolumab to assess overall safety and potential efficacy in a greater number of patients. Patients in the expansion phase of the study may continue treatment up to 18 three-week cycles or until significant disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Nab-Rapamycin; Biological: Nivolumab

INTERVENTIONS:
Drug: Nab-Rapamycin — Escalating doses of ABI-009 will be given IV over 30 min for 2 of every 3 weeks beginning Day 8 Cycle 2. Only nivolumab will be given in Cycle 1. At Dose Level 1, 3-6 patients will receive 56 mg/m^2; at Dose Level 2, 3-6 six patients will receive 75 mg/m^2; and at Dose Level 3, 3-6 patients will receive 100 mg/m^2.
  Other Names: ABI-009
Biological: Nivolumab — A defined dose of nivolumab, 3 mg/kg, will be given IV over 30 minutes q 3 weeks
  Other Names: Opdivo

SUMMARY:
This study investigates the safety/toxicity and potential anti-tumor activity of sequential administration of nivolumab and escalating doses of the mammalian target of rapamycin (mTOR) inhibitor nab-rapamycin (ABI-009) in advanced Ewing's sarcoma, perivascular epithelioid cell tumor (PEComa), epithelioid sarcoma, desmoid tumor, chordoma, non-small cell lung cancer, small cell lung cancer, urothelial carcinoma, melanoma, renal cell carcinoma, squamous cell carcinoma of head and neck, hepatocellular carcinoma, classical Hodgkin's lymphoma, high microsatellite instability (MSI-H)/ mismatch repair deficient (dMMR) metastatic colorectal cancer, and tumors with genetic mutations sensitive to mTOR inhibitors.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the maximum tolerated dose (MTD) of ABI-009, an mTOR inhibitor, when given sequentially with nivolumab in advanced Ewing's sarcoma, PEComa, epithelioid sarcoma, desmoid tumor, chordoma, non-small cell lung cancer, small cell lung cancer, urothelial carcinoma, melanoma, renal cell carcinoma, squamous cell carcinoma of head and neck, hepatocellular carcinoma, classical Hodgkin's lymphoma, MSI-H/dMMR metastatic colorectal cancer, and tumors with genetic mutations sensitive to mTOR inhibitors.

The secondary objectives are to investigate the disease control rate (DCR) and progression free survival (PFS) using nivolumab/ABI-009 combination therapy in advanced Ewing's sarcoma, PEComa, epithelioid sarcoma, desmoid tumor, chordoma, non-small cell lung cancer, small cell lung cancer, urothelial carcinoma, melanoma, renal cell carcinoma, squamous cell carcinoma of head and neck, hepatocellular carcinoma, classical Hodgkin's lymphoma, MSI-H/dMMR metastatic colorectal cancer, and tumors with genetic mutations sensitive to mTOR inhibitors.

The exploratory objectives are (1) To correlate progression free survival (PFS) based on Immune-related Response Criteria (irRECIST) with that based on RECIST v1.1, and (2) To correlate PFS with programmed cell death protein 1 (PD-1) and programmed death-ligand 1 (PD-L1) expression in patients' tumors.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study only if all of the following criteria are met:

1. Patients must have a histologically confirmed diagnosis of Ewing's sarcoma, PEComa, epithelioid sarcoma, desmoid tumor, chordoma, non-small cell lung cancer, small cell lung cancer, urothelial carcinoma, melanoma, renal cell carcinoma, squamous cell carcinoma of head and neck, hepatocellular carcinoma, classical Hodgkin's lymphoma, MSI-H/dMMR metastatic colorectal cancer, and tumors with genetic mutations sensitive to mTOR inhibitors, that is either metastatic or locally advanced and for which surgery is not a recommended option.
2. Patients must have one or more measurable target lesions by CT scan or MRI. Measurable disease by RECIST v1.1.
3. Patients must not have been previously treated with a PD-1 inhibitor in combination with an mTOR inhibitor.
4. Prior treatment (investigational or other), chemotherapy, radiotherapy, surgery, or other therapeutic agents (except immunotherapy and mTOR inhibitors) is allowed, if completed after 5 half-lives or ≥28 days prior to enrollment, whichever is shorter.
5. Eligible patients, 12 years or older, with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. Patients must have the following blood chemistry levels at screening (obtained ≤14 days prior to enrollment (local laboratory):

   1. total bilirubin ≤1.5 x upper limit of normal (ULN) mg/dl
   2. Aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 x ULN if attributable to liver metastases)
   3. serum creatinine ≤1.5 x ULN
7. Adequate biological parameters as demonstrated by the following blood counts at screening (obtained ≤14 days prior to enrollment, local laboratory):

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L;
   2. Platelet count ≥100,000/mm3 (100 × 109/L);
   3. Hemoglobin ≥9 g/dL.
8. Serum triglyceride <300 mg/dL; serum cholesterol < 350 mg/dL.
9. Male or non-pregnant and non-breast feeding female:

   Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting investigational product (IP) and while on study medication and have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. A second form of birth control is required even if she has had a tubal ligation.

   Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study. A second form of birth control is required even if he has undergone a successful vasectomy.
10. Life expectancy of >3 months, as determined by the investigator.
11. Ability to understand and sign informed consent.
12. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Concurrent or prior immunotherapy with a PD-1 inhibitor in combination with an mTOR inhibitor.
2. Known active uncontrolled or symptomatic central nervous system (CNS) metastases. A patient with controlled and asymptomatic CNS metastases may participate in this study. As such, the patient must have completed any prior treatment for CNS metastases ≥28 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
3. Active gastrointestinal bleeding.
4. Pre-existing thyroid abnormality is allowed provided thyroid function can be controlled with medication.
5. Uncontrolled serious medical or psychiatric illness. Patients with a "currently active" second malignancy other than non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pT2 with Gleason Score ≤ 6 and postoperative prostate-specific antigen (PSA) <0.5 ng/mL), or other adequately treated carcinoma-in-situ are ineligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥1 year).
6. Liver-directed therapy within 2 months of enrollment. Prior treatment with radiotherapy (including radio-labeled spheres and/or cyberknife, hepatic arterial embolization (with or without chemotherapy) or cryotherapy/ablation) is allowed if these therapies did not affect the areas of measurable disease being used for this protocol.
7. Recent infection requiring systemic anti-infective treatment that was completed ≤14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
8. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy.
9. Unstable coronary artery disease or myocardial infarction during preceding 6 months.
10. Receiving any concomitant antitumor therapy.
11. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
12. Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfenadine) within the 14 days prior to receiving the first dose of ABI-009.
13. Known Human Immunodeficiency Virus (HIV).
14. Active Hepatitis B or Hepatitis C.
15. Non-oncology vaccine therapy used for prevention of infectious disease within 4 weeks of trial enrollment
16. Autoimmune disease including rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis and motor neuropathy considered to be of autoimmune origin (e.g. Guillain-Barre Syndrome)
17. Systemic immunosuppression, including HIV positive status with or without AIDS
18. Skin rash (psoriasis, eczema) affecting > 25% body surface area
19. Inflammatory bowel disease (Crohn's or ulcerative colitis)
20. Ongoing or uncontrolled diarrhea within 4 weeks of trial enrollment
21. Recent history of acute diverticulitis, intraabdominal abscess or gastrointestinal obstruction within 6 months of trial enrollment, which are known risk factors for bowel perforation
22. Current, active or previous history of heavy alcohol abuse
23. Pituitary endocrinopathy
24. Adrenal insufficiency or excess

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erlinda M Gordon, MD, Principal Investigator — Sarcoma Oncology Research Center
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gonzalez-Angulo AM, Meric-Bernstam F, Chawla S, Falchook G, Hong D, Akcakanat A, Chen H, Naing A, Fu S, Wheler J, Moulder S, Helgason T, Li S, Elias I, Desai N, Kurzrock R. Weekly nab-Rapamycin in patients with advanced nonhematologic malignancies: final results of a phase I trial. Clin Cancer Res. 2013 Oct 1;19(19):5474-84. doi: 10.1158/1078-0432.CCR-12-3110. PMID 24089446
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, single-center, dose-finding phase IB study using a fixed dose of nivolumab and escalating doses of nab-sirolimus given intravenously. Patients were enrolled from August 2017 to July 2021 at the Sarcoma Oncology Center, Santa Monica CA 90403. The study was conducted in accordance with the Declaration of Helsinki and approved by the Western Institutional Review Board (Protocol Code 20151429 on September 8, 2017) for studies involving humans.
Groups:
- Dose Escalation Phase 1 Dose Level I; Dose Escalation Phase 1 Dose Level II; Dose Escalation Phase 1 Dose Level III: The study will employ the standard "cohort of three" design. Three patients are treated at each dose level with expansion to six patients per cohort if DLT is observed in one of the three initially enrolled patients at each dose level. If no DLT occurs after 2 doses, escalation to the next dose level will be permitted. The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced DLT, with the next higher dose level having at least two patients who experienced DLT. Patients in the dose escalation study may continue treatment at their designated dose levels up to eighteen 3-week cycles or until significant disease progression or unacceptable toxicity occurs. No intra-patient dose escalation will take place.
- Expansion Phase 1b Part: Following dose escalation, an additional 22-28 patients will receive ABI-009 at the MTD and defined doses of nivolumab to assess overall safety and potential efficacy in a greater number of patients. Patients in the expansion phase of the study may continue treatment up to 18 3-week treatment cycles or until significant disease progression or unacceptable toxicity occurs.
Period: Overall Study
Arm/Group | Dose Escalation Phase 1 Dose Level I | Dose Escalation Phase 1 Dose Level II | Dose Escalation Phase 1 Dose Level III | Expansion Phase 1b Part
Started | 3 | 3 | 3 | 25
Completed | 3 | 3 | 3 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: 56 mg/m^2; Phase 1: 75mg/m^2; Phase 1: 100 mg/m^2; Phase 1b: 100 mg/m^2: This was an open-label, single-center, dose-finding phase IB study using a fixed dose of nivolumab and escalating doses of nab-sirolimus given intravenously. Patients were enrolled from August 2017 to July 2021. The study was conducted in accordance with the Declaration of Helsinki and approved by the Western Institutional Review Board (Protocol Code 20151429 on September 8, 2017) for studies involving humans.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 56 mg/m^2 | Phase 1: 75mg/m^2 | Phase 1: 100 mg/m^2 | Phase 1b: 100 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 25 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 25 | 31
  >=65 years | 2 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 1 | 2 | 1 | 11 | 15
  Sex: Male | 2 | 1 | 2 | 14 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 22 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of ABI-009
Description: The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced dose-limiting toxicity (DLT), with the next higher dose level having at least two patients who experienced DLT.
Time Frame: Week 6
Population: Intention-to-treat population (all participant assigned to the Phase I dose escalation part of the study).
Measure: Number; unit: mg/m^2
Groups:
- Dose Escalation Phase 1: The study will employ the standard "cohort of three" design. Patients receive ABI-009 in level I dose - 56 mg/m^2, in level II dose - 75 mg/m^2, and level III dose - 100 mg/m^2, each with defined dose of nivolumab - 240 mg IV 30 min. q 3 weeks.
Arm/Group | Dose Escalation Phase 1
Number analyzed (Participants) | 9
mg/m^2 | 100

2. Secondary Outcome: Disease Control Rate
Description: The disease control rate is the percent of patients with complete response, partial response and stable disease.
Time Frame: 12 weeks
Population: Per pre-specified analysis, only participants in the expansion phase of the study were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Expansion Phase 1b: Following dose escalation, an additional 25 patients will receive ABI-009 at the MTD and defined doses of nivolumab to assess overall safety and potential efficacy in a greater number of patients. Patients in the expansion phase of the study may continue treatment up to 18 three-week cycles or until significant disease progression or unacceptable toxicity occurs.
Arm/Group | Expansion Phase 1b
Number analyzed (Participants) | 25
Participants | 22

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is the time from start of treatment to disease progression or death.
Time Frame: 24 weeks
Population: Per pre-specified analysis, only participants in the expansion phase of the study were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase 1b
Number analyzed (Participants) | 25
Participants | 22

4. Secondary Outcome: Overall Survival
Description: The overall survival is the time from treatment initiation to death.
Time Frame: 30 weeks
Population: Per pre-specified analysis, only participants in the expansion phase of the study were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase 1b
Number analyzed (Participants) | 25
Participants | 22

ADVERSE EVENTS:
Time Frame: 3.8 years
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information does not differ from that of the clinicaltrials.gov.
Groups:
- Dose Escalation Phase 1 Part I: The study will employ the standard "cohort of three" design. Patients receive ABI-009 in level I dose - 56 mg/m^2 and defined dose of nivolumab - 240 mg IV 30 min. q 3 weeks.
- Dose Escalation Phase 1 Part II: The study will employ the standard "cohort of three" design. Patients receive ABI-009 in level II dose - 75 mg/m^2 and defined dose of nivolumab - 240 mg IV 30 min. q 3 weeks.
- Dose Escalation Phase 1 Part III: The study will employ the standard "cohort of three" design. Patients receive ABI-009 in level III dose - 100 mg/m^2 and defined dose of nivolumab - 240 mg IV 30 min. q 3 weeks.
Arm/Group | Dose Escalation Phase 1 Part I | Dose Escalation Phase 1 Part II | Dose Escalation Phase 1 Part III | Expansion Phase 1b
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 21/25
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 3/25
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase 1 Part I (N=3) | Dose Escalation Phase 1 Part II (N=3) | Dose Escalation Phase 1 Part III (N=3) | Expansion Phase 1b (N=25)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — One (3.2%) had acute dehydration.
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — Three (9.7%) patients had thrombocytopenia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase 1 Part I (N=3) | Dose Escalation Phase 1 Part II (N=3) | Dose Escalation Phase 1 Part III (N=3) | Expansion Phase 1b (N=25)
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Two patients developed Grade 2 oral mucositis.

LIMITATIONS AND CAVEATS:
The study was completed with a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03190174/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03190174/ICF_001.pdf